CLINICAL TRIAL: NCT00580307
Title: Surgical Correction of Contact Point Headaches - Randomized Controlled Trial. [Rhinogenic Headache Improvement After Nasal Operation] Trial
Brief Title: Rhinogenic Headache Improvement After Nasal Operation
Acronym: RHINO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1089377
Record Dates: First submitted 2007-12-12; First posted 2007-12-24 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Headache
Keywords: Headache; Rhinogenic; Nose; Nasal septum; Deviated septum; Surgery; Septoplasty; Turbinoplasty; Contact point; HIT-6
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septoplasty (Placebo Comparator): Septoplasty only
  Interventions: Procedure: Septoplasty
- Septoplasty and correction (Experimental): Septoplasty and endoscopic contact point correction
  Interventions: Procedure: Septoplasty and endoscopic contact point correction

INTERVENTIONS:
Procedure: Septoplasty — Surgical straightening of nasal septum
  Arms: Septoplasty
Procedure: Septoplasty and endoscopic contact point correction — Septoplasty (as previously described). Contact point correction: structures of the lateral nasal wall that impinge on the nasal septum are mobilized to a more lateral position under endoscopic guidance.
  Other Names: Turbinoplasty
  Arms: Septoplasty and correction

SUMMARY:
Objective: To determine the efficacy of surgical correction of intranasal mucosal contact points in improving quality of life and decreasing medication use in patients with rhinogenic headaches.

DETAILED DESCRIPTION:
Significance: Chronic, debilitating headaches that resist maximal medical treatment by various headache specialists are sometimes linked to structural anomalies within the nose that exert pressure on apposing mucosal surfaces. A number of otolaryngologists have reported success in alleviating rhinogenic headaches with contact point correction surgery. This practice is supported by anecdotal reports along with retrospective and observational studies; however, a prospective study with an appropriate surgical control group has not been conducted. Because the specific effect of contact point correction has not yet been differentiated from the placebo effect of surgery itself, many headache specialists are reluctant to recommend surgical evaluation for their patients. To demonstrate the efficacy of contact point correction surgery to both the headache and otolaryngology communities - and thus, to make this treatment option more widely available to rhinogenic headache sufferers - a randomized controlled trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 2 months) pain or pressure over nasal bridge, glabella, or forehead
* Unilateral or bilateral nasal septal deviation that is chronically symptomatic (e.g. nasal airway obstruction)
* Failure of standard medical therapy for headache
* Symptomatic contact points as demonstrated by physical examination, sinus CT and nasal endoscopy
* Relief of headache after application of topical anesthetic to contact points
* Contact points that remain after mucosal decongestion
* Absence of any other obvious cause of headaches after a thorough evaluation by a neurologist, ophthalmologist, dentist, internist, or other related specialist

Exclusion Criteria:

* Previous sinonasal surgery
* Active acute sinonasal disease:

  1. Seasonal allergic exacerbations with mucosal swelling
  2. Acute infectious rhino-sinusitis
* Chronic sinonasal problems:

  1. Severe nasal polyps mimicking contact points
  2. Mucoceles protruding from sinuses into nasal cavity
  3. Nasal and sinus tumors
* General medical condition that precludes elective surgery (including pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Between-group difference in patient-rated headache improvement at 10 days, 6 weeks, 6 months and 12 months post-intervention, as measured by a validated questionnaire, the Headache Impact Test - 6 (HIT-6™). | 12 months

SECONDARY OUTCOMES:
Between-group differences in subject responses to a non-validated questionnaire so as to permit comparison with previous studies. Additionally, headache medication use will be examined as a secondary end-point. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Page, MD, Principal Investigator — Dept. OtoHNS, U. Missouri - Columbia; Alvis L Barrier, MD, Study Director — Dept. OtoHNS, U. Missouri- Columbia; Karen H Calhoun, MD, FACS, Study Chair — Dept. OtoHNS, U. Missouri - Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided